CLINICAL TRIAL: NCT00858962
Title: A Study of the Pharmacokinetic and Pharmacodynamic Interactions Between Raltegravir (Isentress) and Buprenorphine
Brief Title: Buprenorphine/Raltegravir Pharmacokinetic Interaction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, R. Douglas Bruce, MD, MA, Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0811004456; R01DA025932 (NIH)
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infection; HIV Infections
Keywords: HIV; Pharmacokinetics; Pharmacodynamics; Buprenorphine; Raltegravir; HIV seronegativity; Interaction
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bup/Ral (Experimental): Buprenorphine and Raltegravir co-administration
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400 mg of raltegravir orally twice daily together with normally prescribed stable dose of buprenorphine for a minimum of 4 days and up to 14 days.
  Other Names: Isentress

SUMMARY:
The main purpose of this protocol is to study the effect of an HIV medication known as Raltegravir on Buprenorphine in people who have been receiving the same dose of Buprenorphine for at least 3 weeks before study entry. This will be determined by giving Raltegravir along with Buprenorphine and by measuring the amount of Raltegravir and Buprenorphine in the blood. The investigators will also learn about the effects of Buprenorphine on Raltegravir and about the safety of taking these two medications together.

DETAILED DESCRIPTION:
A large number of people who are infected with HIV have acquired it through injection drug use. Some of these people are currently being treated with Buprenorphine for their addiction and with medications for HIV infection. Raltegravir is a medication that was approved by the Food and Drug Administration (FDA) for the treatment of HIV infection. Raltegravir acts by making it more difficult for the virus that causes AIDS to multiply and cause more damage to the immune system in someone who is HIV infected.

Earlier studies looking at the effect of Buprenorphine and HIV medications have shown that Buprenorphine and some HIV medications act differently when taken together. It is important to learn if taking Buprenorphine and HIV medications together results in changes in the blood level of either medication. If the HIV medication affects the level of Buprenorphine in the blood, an individual taking Buprenorphine and HIV medications may experience symptoms of withdrawal, even while taking their usual dose of Buprenorphine. On the other hand, if Buprenorphine decreases the amount of HIV medication in the blood, then the HIV medication may be less effective in controlling HIV infection. It is therefore important to learn if Raltegravir and Buprenorphine will affect each other when taken together.

In order to learn about the effects of Buprenorphine and Raltegravir, we will need to measure the amount of Buprenorphine in your blood for 24 hours before you have taken Raltegravir and then compare that to the amount of Buprenorphine in your blood after you have taken Buprenorphine and Raltegravir together .

ELIGIBILITY:
Inclusion Criteria:

* Patients who are opioid dependent on long-term buprenorphine/naloxone (BUP/NLX) maintenance (minimum of 4 weeks) and who must remain at a stable dose of buprenorphine for at least 3 weeks deemed by the investigator to have acceptable medical history, physical examination and clinical laboratory evaluations consistent with BUP maintenance will be eligible to participate in the study.
* Body weight >60 kg for males and >40 kg for females
* Male or females, ages > 21 to < 60 years.
* Women of childbearing potential (WOCBP) must not be nursing or pregnant and must be on adequate non-hormonal contraception to avoid pregnancy. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Study Day 1.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks before and after the study.
* Use of an oral, injectable or implantable hormonal contraceptive agent within 3 months of enrollment and throughout the study.
* Women who are currently pregnant or breastfeeding.
* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* Proven or suspected acute hepatitis at the time of study entry
* Any major surgery within 4 weeks of enrollment. Minor surgical procedures requiring local anesthesia are exceptions.
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of enrollment.
* Blood transfusion within 4 weeks of enrollment.
* Inability to tolerate oral medication.
* Inability to tolerate venipuncture and/or absence of secure venous access.
* Inability to refrain from smoking during in-residence period
* Evidence of organ dysfunction or any clinically relevant (as determined by the investigator) deviations from the norms observed in a buprenorphine/naloxone treated population in physical examination, vital signs, or clinical laboratory determinations.
* Positive breathalyzer alcohol test, or positive urine screen for barbiturates, benzodiazepines, amphetamines, cocaine or opioids other than buprenorphine/naloxone.
* Subjects with AST, ALT or bilirubin > 3.0X the upper limit of normal
* Hemoglobin < 9 g/dL, and platelet count < 75,000/mm3.
* Positive serum or urine for HCG.
* History of any significant drug allergy, drug rash or sensitivity to any class of drugs relevant to the study drugs.
* HIV antibody positive
* Exposure to any investigational drug within 4 weeks of enrollment and throughout the study.
* Prior exposure to Raltegravir.
* Use of any agent (prescribed or otherwise) within 2 weeks of dosing, that is known or suspected to induce or inhibit drug metabolizing enzymes (e.g., cimetidine and compounds in the barbiturate and phenothiazine classes), affect renal tubular secretion (e.g., probenecid, beta-lactam antibiotics), gastrointestinal motility (e.g., metoclopramide, propantheline, loperamide, or narcotic analgesics or opioids other than buprenorphine/naloxone), or uric acid metabolism (e.g., allopurinol) or gastrointestinal pH (including antacids, H2-receptor antagonists, proton pump inhibitors etc.).
* Use of over-the-counter medications and herbal preparations, within 1 week prior to enrollment and throughout the study.
* Use of St. John's Wort (Hypericum) within four weeks prior to study enrollment and throughout the study.
* Consumption of grapefruit or grapefruit juice within 1 week of study entry and throughout the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Bruce, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir (400mg Twice Per Day): Subjects were maintained on Buprenorphine/Naloxone (BUP/NLX) for 3 weeks prior to Raltegravir administration to achieve steady state during baseline. Subsequently, subjects were co-administered raltegravir (400mg twice per day)and BUP/NLX. All subjects received 16/4 mg of BUP/NLX daily, except for 1 patient who received 32/8 mg daily.
Period: Overall Study
Arm/Group | Raltegravir (400mg Twice Per Day)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir (400mg Twice Per Day)
Number analyzed (Participants) | 12
Age Continuous [Mean (Full Range); unit: years] | 44 [30 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of BUP/NLX With Raltegravir (hr*ng/mL)
Description: PK parameters of BUP were determined by non-compartmental methods. AUC of BUP was determined by use of the trapezoidal rule.
Time Frame: 6-14 days after beginning co-administration of drugs
Population: All subjects who completed study were included in the analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Raltegravir (400mg Twice Per Day)
Number analyzed (Participants) | 12
hr*ng/mL | 56.0 (17.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of each subject's participation in the study.
Groups:
- Bup/Ral: HIV negative subjects currently enrolled in Buprenorphine maintenance therapy on a stable dose of BUP for at least 3 weeks were admitted to the HRU for PK sampling at intervals over a 24 hour period. Subjects then received RAL and BUP co-administration for a minimum of 4 days after which a second series of blood draws at intervals over a 24 hour period were conducted.
Arm/Group | Bup/Ral
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
The sample size was small, though within the range of similar drug-drug interaction studies. This study utilized a within-subject design with patients acting as their own controls (thereby resulting in less intra-patient variability).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less